CLINICAL TRIAL: NCT00112827
Title: Tandem High-Dose Therapy With Melphalan and Total Marrow Irradiation (TMI) With Peripheral Blood Progenitor Cell Support and Lenalidomide Maintenance in Multiple Myeloma: A Phase I/II Trial
Brief Title: Melphalan and Radiation Therapy Followed By Lenalidomide in Treating Patients Who Are Undergoing Autologous Stem Cell Transplant for Stage I, Stage II, or Stage III Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 04064; CDR0000428410 (Other: NCI PDQ)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Refractory Multiple Myeloma; Smoldering Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Melphalan; Peripheral Blood Stem Cell Transplantation; Filgrastim; Granulocyte Colony-Stimulating Factor; In Situ Hybridization, Fluorescence; Cytogenetic Analysis; Cyclophosphamide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): See Detailed Description
  Interventions: Radiation: total marrow irradiation; Drug: melphalan; Procedure: peripheral blood stem cell transplantation; Biological: filgrastim; Genetic: fluorescence in situ hybridization; Genetic: cytogenetic analysis; Drug: cyclophosphamide; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation; Drug: lenalidomide

INTERVENTIONS:
Radiation: total marrow irradiation — Undergo irradiation
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin; Melfalan
Procedure: peripheral blood stem cell transplantation — Undergo transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Biological: filgrastim — Given IV
  Other Names: G-CSF; granulocyte colony-stimulating factor; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor
Genetic: fluorescence in situ hybridization — Correlative studies
  Other Names: fluorescence in situ hybridization (FISH)
Genetic: cytogenetic analysis — Correlative studies
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Procedure: autologous-autologous tandem hematopoietic stem cell transplantation — Undergo transplantation
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid

SUMMARY:
RATIONALE: Melphalan, a chemotherapeutic agent, has been found to be an effective treatment choice for destroying myeloma cells, especially when given at high (bone marrow ablative) doses. Total marrow irradiation (TMI)/ablative dose radiation therapy is another modality capable of destroying myeloma cells. Autologous peripheral blood/stem cell transplant (ASCT) given after either melphalan or following TMI (aimed at the bone marrow containing areas of the skeleton, the site of origin of myeloma cells) will shorten the duration/alleviate the severity of both melphalan and marrow irradiation-associated side effects. Lenalidomide, an effective agent on its own right for the treatment of myeloma, has been shown to further enhance the beneficial effects of autologous stem cell transplants when given as maintenance therapy.

PURPOSE: This previously phase I trial established the maximum tolerated dose of TMI at 1600 cGy. The phase II part of this study is ongoing and is studying the effects of high-dose melphalan and ASCT, followed by TMI and a second ASCT, with subsequent maintenance lenalidomide. The study is conducted in patients with stages I-III myeloma, with specific emphasis on assessing complete and very good partial response rate conversions, progression-free and overall survival, and safety/feasibility of delivering the planned treatment regimen.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and toxicities of tandem cycle ablative therapy consisting first of high-dose melphalan and then escalating doses of fractionated total marrow irradiation (TMI) using helical tomotherapy in patients with advanced multiple myeloma.

II. To establish the maximum tolerated dose of TMI using helical tomotherapy. III. To assess response rate, progression free and over-all survival following treatment with tandem cycle ablative therapy consisting first of high-dose melphalan and then escalating doses of TMI using helical tomotherapy with Dexamethasone/Thalidomide maintenance therapy in patients with advanced multiple myeloma.

IV. To assess the feasibility of adding decadron and thalidomide as maintenance following the second cycle of high-dose therapy.

SECONDARY OBJECTIVES:

I. To perform cytogenetic, gene rearrangement, and fluorescence in situ hybridization (FISH) studies on baseline and post-treatment bone marrow and blood specimens and correlate the presence/persistence of these features with treatment outcome.

II. To bank/develop cell lines developed for future investigations of tumor biology, and for potential assessment of efficacy of novel therapeutic agents.

OUTLINE: This is a dose-escalation study of total marrow irradiation (TMI).

PRIMING AND APHERESIS: Patients receive cyclophosphamide IV over 2 hours. Patients also receive filgrastim IV or subcutaneously daily beginning 24 hours after the administration of cyclophosphamide and continuing until apheresis is complete. Patients undergo apheresis until an adequate number of peripheral blood stem cells are collected.

ABLATIVE THERAPY:

Course 1: Patients receive high-dose melphalan IV over 30 minutes on days -2 and -1. Patients then undergo autologous PBSC transplantation on day 0 and receive filgrastim IV or subcutaneously beginning on day 5 and continuing until blood counts recover.

Course 2: Beginning 6-18 weeks later, patients undergo TMI once or twice daily on days -4 to -1. Patients then undergo autologous peripheral blood stem cell transplant and receive filgrastim IV or subcutaneously beginning on day 5 and continuing until blood counts recover.

MAINTENANCE THERAPY: Beginning within 6-8 weeks of day 0 of course 2 (TMI), patients receive oral lenalidomide daily. Courses repeat every 28 days for approximately 3 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days, every 6 months for 1 year, and then annually for at least 2 years.

ELIGIBILITY:
Criteria

* Patients with multiple myeloma (stages I-III) will be eligible if they are either in response, or have stable disease
* Patients with smoldering myeloma are eligible if there is evidence of progressive disease requiring therapy (>= 25% increase in M protein levels or Bence Jones excretion; Hgb =< 10.5 g/dl; frequent infections; hypercalcemia; rise in serum creatinine above normal on two separate occasion)
* Patients with non-quantifiable monoclonal proteins are eligible provided they meet other criteria for multiple myeloma, or smoldering myeloma, and they have evaluable or measurable disease by other (radiographic) means
* Unlimited prior chemotherapy regimens allowed
* KPS >= 70%
* Patients with Waldenstrom's macroglobulinemia are not eligible
* Less than 18 months since diagnosis
* No contraindication to the collection of a minimum of 4 x 10^6 CD34+ cells/kg by apheresis
* All patients must have signed a voluntary, informed consent in accordance with institutional and federal guidelines
* Adequate hepatic function as demonstrated by bilirubin, =< 1.5 mg/dl, and SGOT and SGPT < 2.5 x upper limits of normal
* Adequate renal function as demonstrated by: creatinine of measured or calculated creatinine clearance of > 50 cc/min
* Absolute neutrophil count of > 1000/ul, platelet count of > 100,000/ul
* Cardiac ejection fraction >= 50% by MUGA scan and/or by echocardiogram
* Adequate pulmonary function as demonstrated by FEV1 > 60% and DLCO > 50% of predicted lower limit
* Hepatitis B antigen, Hepatitis C RNA and HIV antibody tests negative
* No other medical, or psychosocial problems, which in the opinion of the primary physician or principal investigator would place the patient at unacceptably high risk from this treatment regimen
* Females of reproductive age not using adequate birth control measures/ or who are pregnant are not eligible
* History of other malignancies within the last 3 years, as long as patients have remained in complete remission for at least 2 years, except for non-melanoma skin cancer and in situ carcinoma of the cervix
* Patients should have finished their prior chemotherapy at least 14 days prior to cyclophosphamide priming, and should have received their last dose of thalidomide, dexamethasone, or bisphosphonate > 10 days prior to cyclophosphamide priming
* Pre-treatment tests must have been performed within 6 weeks prior to initiation of cyclophosphamide; A CBC, platelet count and comprehensive chemistry panel should be performed within 1 week prior to initiating cyclophosphamide priming
* Known hypersensitivity to Filgrastim or to E. coli derived proteins is an exclusion
* Inability to lie supine in a full body cast for approximately 30 minutes, the anticipated duration of each treatment session, is an exclusion
* Previous radiation therapy to more than 20% of bone marrow containing areas, or to any area exceeding 2000 cGy, is an exclusion
* Patients must be fully aware of the teratogenic potential of thalidomide and agree to fully comply with the mandated guidelines regarding contraception as stated in the informed consent and the patient warning document attached to the consent form
* Women of childbearing potential must have a negative pregnancy test performed within 24 hours prior to beginning thalidomide, except for woman who have been postmenopausal for at least 2 years, or underwent hysterectomy
* Use of effective means of contraceptive should be started at least 2 weeks prior to initiating thalidomide

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Cohort 1 (Total TMI Dose: 1000 cGy); Phase 1 Cohort 2 (Total TMI Dose: 1200 cGy); Phase 1 Cohort 3 (Total TMI Dose: 1400 cGy); Phase 1 Cohort 4 & Phase 2 MTD (Total TMI Dose:1600 cGy); Phase 1 Cohort 5 (Total TMI Dose: 1800 cGy): See Detailed Description
  total marrow irradiation: Undergo irradiation escalating according to the following schedule 1000cGy, 1200cGy, 1400cGy, 1600cGy, 1800cGy
  melphalan: Given IV
  peripheral blood stem cell transplantation: Undergo transplantation
  filgrastim: Given IV
  fluorescence in situ hybridization: Correlative studies
  cytogenetic analysis: Correlative studies
  cyclophosphamide: Given IV
  autologous-autologous tandem hematopoietic stem cell transplantation: Undergo transplantation
  lenalidomide: Given orally
Period: Overall Study
Arm/Group | Phase 1 Cohort 1 (Total TMI Dose: 1000 cGy) | Phase 1 Cohort 2 (Total TMI Dose: 1200 cGy) | Phase 1 Cohort 3 (Total TMI Dose: 1400 cGy) | Phase 1 Cohort 4 & Phase 2 MTD (Total TMI Dose:1600 cGy) | Phase 1 Cohort 5 (Total TMI Dose: 1800 cGy)
Started | 3 | 4 | 4 | 36 | 7
Completed | 3 | 4 | 4 | 36 | 7
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Cohort 1 (Total TMI Dose: 1000 cGy) | Phase 1 Cohort 2 (Total TMI Dose: 1200 cGy) | Phase 1 Cohort 3 (Total TMI Dose: 1400 cGy) | Phase 1 Cohort 4 & Phase 2 MTD (Total TMI Dose:1600 cGy) | Phase 1 Cohort 5 (Total TMI Dose: 1800 cGy) | Total
Number analyzed (Participants) | 3 | 4 | 4 | 36 | 7 | 54
Age, Continuous [Median (Full Range); unit: years] | 49 [42 to 53] | 56 [53 to 66] | 54 [52 to 62] | 54 [31 to 67] | 54 [36 to 64] | 54 [31 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 13 | 4 | 23
  Male | 2 | 2 | 1 | 23 | 3 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0 | 0 | 0 | 6 | 2 | 8
  Caucasian | 3 | 2 | 4 | 22 | 4 | 35
  Hispanic | 0 | 1 | 0 | 5 | 1 | 7
  Asian | 0 | 1 | 0 | 2 | 0 | 3
  Other | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 4 | 36 | 7 | 54

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The highest dose tested (Total Marrow Irradiation) in which there is no treatment related mortality and none or only one patient experienced dose limited toxicity (DLT) attributable to the study drug(s), when at least six were fully treated at that dose and fully followed for toxicity. The MTD is one dose level below the lowest dose tested in which 2 or more patients experienced DLT attributable to the treatment or there was a treatment related death. At least 6 patients will be treated at the MTD.
Time Frame: 8 weeks from start of treatment, up to 2 years
Population: All patients enrolled in the dose-finding portion of the study.
Measure: Number; unit: cGy
Groups:
- Treatment Arm: See Detailed Description
  total marrow irradiation: Undergo irradiation escalating according to the following schedule 1000cGy, 1200cGy, 1400cGy, 1600cGy, 1800cGy
  melphalan: Given IV
  peripheral blood stem cell transplantation: Undergo transplantation
  filgrastim: Given IV
  fluorescence in situ hybridization: Correlative studies
  cytogenetic analysis: Correlative studies
  cyclophosphamide: Given IV
  autologous-autologous tandem hematopoietic stem cell transplantation: Undergo transplantation
  lenalidomide: Given orally
Arm/Group | Treatment Arm
Number analyzed (Participants) | 24
cGy | 1600

2. Primary Outcome: Number of Subjects With Response
Description: Response defined as complete response or very good partial response. Complete response defined as the absence of bone marrow or blood findings of multiple myeloma on at least 2 measurements at a minimum of a 6 week interval. Thus all evidence of serum and urinary M-components must disappear on electrophoresis as well as by immunofixation studies. The follow-up bone marrow may not contain more than 5% plasma cells on aspiration or core biopsy and no evidence of increasing anemia. Skeletal X-rays must either show recalcification or no change in osteolytic lesions. Resolution of soft tissue plasmocytomas. Very good partial response defined as reduction of bone marrow or blood findings of multiple myeloma on at least 2 measurements at a minimum of a 6 week interval by greater than or equal to 90%.
Time Frame: Evaluated after each course until completion of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1 (Total TMI Dose: 1000 cGy) | Phase 1 Cohort 2 (Total TMI Dose: 1200 cGy) | Phase 1 Cohort 3 (Total TMI Dose: 1400 cGy) | Phase 1 Cohort 4 & Phase 2 MTD (Total TMI Dose:1600 cGy) | Phase 1 Cohort 5 (Total TMI Dose: 1800 cGy)
Number analyzed (Participants) | 3 | 4 | 4 | 36 | 7
Participants | 3 | 3 | 2 | 20 | 4

3. Primary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Event defined as death due to any cause.
Time Frame: From date of treatment until the date of death from any cause, assessed up to 14 years
Population: Overall survival was calculated for aggregated arms, due to small number of patients in most treatment arms.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 54
months | 95.8 [52.4 to NA] — Upper 95% confidence interval was not reached.

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 14 years and 3 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Phase 1 Cohort 1 (Total TMI Dose: 1000 cGy) | Phase 1 Cohort 2 (Total TMI Dose: 1200 cGy) | Phase 1 Cohort 3 (Total TMI Dose: 1400 cGy) | Phase 1 Cohort 4 & Phase 2 MTD (Total TMI Dose:1600 cGy) | Phase 1 Cohort 5 (Total TMI Dose: 1800 cGy)
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/4 | 4/4 | 20/36 | 4/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4 | 6/36 | 3/7
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/4 | 33/36 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1 (Total TMI Dose: 1000 cGy) (N=3) | Phase 1 Cohort 2 (Total TMI Dose: 1200 cGy) (N=4) | Phase 1 Cohort 3 (Total TMI Dose: 1400 cGy) (N=4) | Phase 1 Cohort 4 & Phase 2 MTD (Total TMI Dose:1600 cGy) (N=36) | Phase 1 Cohort 5 (Total TMI Dose: 1800 cGy) (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1 (Total TMI Dose: 1000 cGy) (N=3) | Phase 1 Cohort 2 (Total TMI Dose: 1200 cGy) (N=4) | Phase 1 Cohort 3 (Total TMI Dose: 1400 cGy) (N=4) | Phase 1 Cohort 4 & Phase 2 MTD (Total TMI Dose:1600 cGy) (N=36) | Phase 1 Cohort 5 (Total TMI Dose: 1800 cGy) (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 1 (1) | 11 (11) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (7) | 4 (10) | 3 (6) | 32 (85) | 7 (28)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mobitz type I (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flashing vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 10 (12) | 5 (5)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5) | 18 (26) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 4 (6) | 2 (3) | 30 (39) | 6 (12)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 6 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 12 (15) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 11 (14) | 0 (0)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastric mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (3)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2) | 7 (9) | 4 (6)
Nausea (Gastrointestinal disorders) | 3 (6) | 4 (7) | 3 (6) | 29 (50) | 7 (15)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 3 (5) | 2 (3) | 23 (32) | 6 (9)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 2 (2) | 1 (2) | 7 (7) | 2 (2)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Edema limbs (General disorders) | 2 (5) | 2 (2) | 1 (1) | 10 (12) | 4 (6)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (8) | 1 (1) | 3 (5) | 26 (48) | 6 (10)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 9 (9) | 1 (1)
General symptom (General disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 1 (1) | 0 (0) | 7 (12) | 5 (5)
Visceral edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune system disorder (Immune system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 4 (6) | 2 (5) | 19 (29) | 7 (13)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 3 (4) | 3 (6) | 17 (27) | 6 (11)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood gonadotrophin abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 5 (8) | 2 (2)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercholesterolemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Leukocyte count decreased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 30 (63) | 4 (11)
Leukopenia (Investigations) | 3 (6) | 4 (13) | 3 (6) | 3 (13) | 3 (37)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 19 (31) | 2 (5)
Lymphopenia (Investigations) | 3 (6) | 4 (11) | 3 (6) | 3 (9) | 3 (23)
Neutrophil count decreased (Investigations) | 3 (6) | 3 (9) | 3 (5) | 28 (57) | 7 (27)
Platelet count decreased (Investigations) | 3 (6) | 4 (10) | 3 (6) | 32 (70) | 7 (43)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (2) | 8 (10) | 3 (3)
Weight loss (Investigations) | 0 (0) | 2 (2) | 0 (0) | 10 (13) | 1 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 21 (32) | 7 (11)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 5 (5) | 3 (7)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 22 (31) | 2 (4)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 3 (4) | 2 (2) | 3 (3) | 3 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5) | 4 (10) | 3 (5) | 3 (8) | 3 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (6) | 4 (8) | 3 (6) | 3 (6) | 3 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 3 (4) | 1 (2) | 3 (5) | 3 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 3 (4) | 1 (2) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 2 (2) | 3 (5) | 3 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 4 (8) | 2 (3) | 3 (7) | 3 (8)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 29 (53) | 4 (10)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 28 (50) | 4 (7)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 2 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 11 (12) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (15) | 3 (4)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 21 (32) | 4 (5)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 18 (28) | 4 (8)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 21 (34) | 4 (7)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (7) | 1 (1) | 0 (0) | 18 (29) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (3) | 10 (13) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 7 (9) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 14 (19) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 5 (5)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (2) | 18 (23) | 3 (4)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4) | 0 (0) | 3 (6) | 21 (35) | 3 (7)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0) | 1 (1) | 10 (11) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4) | 1 (2) | 1 (1) | 11 (16) | 4 (5)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 11 (15) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 1 (1)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 22 (29) | 6 (9)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (7) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 1 (2)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 9 (12) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT00112827/Prot_SAP_000.pdf